CLINICAL TRIAL: NCT06156098
Title: Bedside Renal Ultrasound Assessment in Critically Ill Patients With Acute Kidney Injury: an Observational Study
Brief Title: Bedside Renal Ultrasound Assessment in Patients With Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202308105
Record Dates: First submitted 2023-10-06; First posted 2023-12-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness
Keywords: Critical Illness; Ultrasound Therapy; Kidney injury
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Exploring the predictive and evaluative value of various indicators of bedside critical renal ultrasound in critically ill patients with acute kidney injury (AKI)

DETAILED DESCRIPTION:
This study aims to perform bedside renal ultrasound examinations on critically ill patients admitted to the ICU (including sepsis, respiratory failure, shock, multiple trauma, etc.) and prospectively observe the relationship between ultrasound parameters and the occurrence and progression of AKI, in conjunction with traditional renal function indicators. This will provide clinicians with a rapid, non-invasive, and visual examination tool at the bedside for early diagnosis and treatment of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 70 years
* Criteria for sepsis patients

Exclusion Criteria:

* Pregnant women.
* Patients with malignant tumors, severe heart failure, chronic renal insufficiency, end stage renal disease, kidney transplantation.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Criteria for sepsis patients: Clear infection focus, Sequential Organ Failure Assessment (SOFA) score ≥ 2. Criteria for septic shock patients: Despite active fluid resuscitation, patients still require vasoactive drugs to maintain blood pressure, with arterial blood lactate level ≥ 2mmol/L. Other critically ill patients include those with shock of various causes,
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Survival | 28 days
  28-day mortality rate

SECONDARY OUTCOMES:
AKI | 28 days
  duration of continuous renal replacement therapy (CRRT)during hospitalization, length of hospital stay, duration of ICU stay, hospital mortality rate, 28-day mortality rate, and other relevant data.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China